CLINICAL TRIAL: NCT03112382
Title: Effect of SLC30A8 rs13266634 Genetic Polymorphism on Zinc Supplementation and Glycemic Control in Egyptian Patients With Type 2 Diabetes Mellitus
Acronym: SLC30A8
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Said, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CL (1461)
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vitamin A; vitamin A, vitamin E drug combination

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- zinc supplement plus vitamin A and E (Active Comparator): patients will be receiving zinc supplement plus vitamin A and E for 3 months.
  Interventions: Drug: zinc supplement plus vitamin A and E
- vitamin A and E (Active Comparator): patients will be receiving equivalent dose of vitamin A and E only for 3 months
  Interventions: Drug: vitamin A and E
- no vitamins (No Intervention): patients will be observed for 3 months

INTERVENTIONS:
Drug: zinc supplement plus vitamin A and E
  Arms: zinc supplement plus vitamin A and E
Drug: vitamin A and E
  Arms: vitamin A and E

SUMMARY:
Study whether SLC30A8 rs13266634 polymorphism is associated with type 2 diabetes mellitus (T2DM) susceptibility in Egyptian patients and study effect of Zn supplementation on glycemic control in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 2 diabetes mellitus.
* Age between 20 and 64 years.
* BMI < 40 kg/m2.
* On fixed oral hypoglycemic dosage for at least 3 months.
* Normal serum creatinine (0.5 to 1.3 mg/dL) with no clinical evidence suggestive kidney disease.
* Normal liver function tests (ALT 7 to 55 U/L, and albumin ˃ 3.5 g/dL).

Exclusion Criteria:

* Those diagnosed of osteomalacia, chronic alcoholics. Patients with type 1 Diabetes Mellitus.
* Those who were taking multivitamin containing zinc or magnesium or any sort of mineral supplements in the previous three months or hormone replacement therapy (estrogen, progesterone) or chelating therapy such as penicillamine, or anticonvulsant (phenytoin, valproate).
* Those with a history of recent surgery or with concurrent acute illness including infectious disease, trauma, inflammatory bowel disease, malignancy, and active immunological diseases, using corticosteroids.
* Pregnant or intend to be pregnant for t least 3 months or lactating women.
* Those who were receiving insulin preparations as a part of diabetes management.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
SLC30A8 rs13266634 polymorphism | one year
  genetic screening of SLC30A8 : solute carrier family 30 member 8
serum zinc | at base line

SECONDARY OUTCOMES:
change from baseline in fasting and 2hr post prandial blood glucose at three months | at base line and after three months
change from baseline in HbA1c at three months | base line and three months
change from baseline in lipid profile at three months | base line and three months
  lipid profile: total cholesterol, triglyceride, HDL, LDL.
change from baseline in fasting serum insulin at three months | baseline and three months
change from baseline in ALT level at three months | baseline and three months
serum Mg | baseline
creatinine level | baseline
serum Iron | baseline
change from baseline in total serum Calcium at three months | baseline and three months

CONTACTS AND LOCATIONS:
Locations (1):
- theoutpatient clinics, department of internal medicine, Cairo University teaching hospitals,, Cairo, Egypt